CLINICAL TRIAL: NCT04192708
Title: Study of Analgesic Efficacy of Different Kinds of Nerve Blocks on Otoplastic Surgery
Brief Title: Study of Analgesic Efficacy of Nerve Blocks on Otoplastic Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Xiao Hu, The attentding physician of Department of Anesthesiology, Eye & ENT Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: chevalier
Record Dates: First submitted 2019-11-25; First posted 2019-12-10 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Microtia; Microtia, Congenital
Keywords: intercostal nerve blocks; ultrasound guidance; thoracic paravertebral block; pain management
MeSH Terms: conditions — Congenital Microtia; Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DV-ICNB group (Experimental): intercostal nerve block under direct vision
  Interventions: Procedure: intercostal nerve block under direct vision
- UG-ICNB group (Experimental): intercostal nerve block under ultrasound guidance
  Interventions: Procedure: intercostal nerve block under ultrasound guidance
- PV group (Experimental): thoracic paravertebral block under ultrasound guidance
  Interventions: Procedure: paravertebral block under ultrasound guidance

INTERVENTIONS:
Procedure: intercostal nerve block under direct vision — When the intercostal nerve is adequated exposed，a surgeon use a 5ml syringe to perform the block and the needle is tilted 15 degree cephalad and advanced towards the caudal rim of the lib，and penetration depth is about 5mm.Then 1% lidocaine and 1/200000 epinephrine 3ml will be injected when negative aspiration of gas or blood.Same procedure will be repeted in the other two exposed intercostal spaces.
  Arms: DV-ICNB group
Procedure: intercostal nerve block under ultrasound guidance — After induction ，an ultrasonographic probe (M-Turbo with the L25 transducer; SonoSite Inc.) is used to scan laterally from the midaxillary line to identify the required anatomic landmarks, while the patients are in a lateral decubitus position. The ribs are identified as hyperechoic streaks, while the pleura appeared as hyperechoic lines between and below the ribs.The needle was advanced towards the caudal rim of the rib until the distal tip is just between the innermost and inner intercostal muscle.1% lidocaine and 1/200000 epinephrine 3ml will be injected when negative aspiration of gas or blood.Same procedure will be repeted in the other two exposed intercostal spaces.
  Arms: UG-ICNB group
Procedure: paravertebral block under ultrasound guidance — Paravertebral block is performed between the thoracic segments T7-8,A linear ultrasound transducer (M-Turbo with the L25×transducer; SonoSite Inc.) is placed to parallel the T7 transverse process so as to identify the T7 spinous process，the T7 transverse process and 7th lib.Then move the probe caudally until the thoracic paravertebral space (TPVS) which is bounded by transverse process,pleura and internal intercostal membrane.Using in-plane technique, we advance the 20-gauge needle(Becton Dickinson Infusion Therapy Sysstems Inc.Sandy,Utah 84070,USA.1.88"，1.1×48mm) until the needle tip penetrates the internal intercostal membrane,9ml mixture of 1% lidocaine and 1/200000 epinephrine after no blood or gas is aspirated.Both PVB and ultrasound-guided ICNB is performed by the same anesthesiologist
  Arms: PV group

SUMMARY:
Background: Children with microtia complain of severe postoperative pain during early postoperative days after rib cartilage harvest for auricular reconstruction. The purpose of this study was to compare the analgesic efficacy of intercostal nerve block (ICNB) and paravertebral block(PV) for preventing postoperative pain after rib cartilage graft for auricular reconstruction in children with microtia.

Methods: In this prospective randomized study, 144 children will be enrolled in this study and randomized into 3 groups:48 patients will received ultrasound-guided ICNB(UG-ICNB group);48 patients will receive ICNB under direct vision (DV-ICNB group) and 48 patients will receive paravertebral block(PV group) undergoing postoperative pain control using either preventive ICNB followed by catheter-based infusion (33 patients, study group) or intravenous (IV) analgesia alone (33 patients, control group). ICNB will be performed by injecting 1% lidocaine plus 1/200000 epinephrine 3ml into each of three intercostal spaces before perichondrial dissection. PV will be carried out by injecting 1% lidocaine plus 1/200000 epinephrine 9ml into T7 paravertebral space just after induction of anesthesia.before wound closure.Each patient receive patient-controlled intravenous analgesia(PCIA) after surgery.Severity of pain,nausea,vomiting and other side effects would be assessed for the postoperative period of 48 hours.

DETAILED DESCRIPTION:
Patients are randomly allocated to one of three groups: receiving intercostal nerve block under direct vision (DV-ICNB group) or receiving intercostal nerve block under ultrasound guidance (UG-ICNB group) or receiving thoracic paravertebral block (PV group) with a block of 6 and 1:1 allocation ratio. . Enrolment and data collection are performed by trained research staff who are not involved in the care of the patients. The treating clinicians are not blinded to the assignment group, but all other staff involved in both the collection and assessment of data are blinded to group allocation.

The primary outcomes is the pain severity,intraoperative fentanyl consumption ,patient-controlled intravenous analgesia(PCIA) requirement and severity of nausea and vomiting during the period of postoperative 48 hours. The secondary outcomes are blood loss during harvesting rib cartilage,fentanyl consumption in post-anaesthesia care unit (PACU),time from PACU arrival to first obtainable pain score,first time of urination,duration of PACU stay and postoperative adverse events such as respiratory depression(defined as respiratory rate <8bpm, requirement of naloxone, and/or peripheral oxygen saturation <90%),pneumothorax and pruritus.

Based on our previous clinical observation, 2.7(SD 0.5)μg/kg of fentanyl is required in DV-ICNB group.We suppose that the requirement could be reduce by 0.3μg/kg in UG-ICNB and PV group .Thus,42 patients are required to detect a significant difference among the groups at a significance level of 95% and a power of 80%. 20 patients were finally enrolled in the study due to possible dropouts (20%).

The continuous variables were expressed as means ± standard deviation (SD) whereas categorical variables were expressed as frequency and percentage for data description. Continous data with a normal distribution is manifested as mean±SD and assessed by Unpaired sample t-test ;continous data with skewed distribution is presented as median(interquartile range,IQR) and assessed by Man-Whitney U test ;categorical data are presented as number and assessed by Chi-square/Fisher exact test. The VAS scores,PCIA consumption and severity of nausea and vomiting of the three groups at multiple time points were analyzed via two-way repeated-measures Anova .

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of microtia
2. Scheduled for rib cartilage harvest from three ribs for auricular reconstruction.

Exclusion Criteria:

1. Requirement for additional surgery
2. Rib cartilage harvest from more or less than three ribs
3. History of analgesic administration (eg, opioids, acetaminophen, or 4.Nonsteroidal anti-inflammatory drugs) 24 hours before premedication

5.History of coagulation disorders or allergy to local anesthetics 6.History of renal insufficiency or an American Society of Anesthesiologists (ASA) physical status that was higher than II 7.Inability to express pain scores or severity of nausea 8.Inability to understand PCIA device use 9.Parental objection to ICNBs or paravertebral block.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Estimated)
Dates: Start 2020-02-17 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Chest pain at rest | Time1:0 minute after the first pain score could be obtained from the patient
  Assessed by Visual Analogue Scale（VAS）,(0,no pain；10，the worst pain)
Chest pain at rest | Time2: 3 hours after surgery
  Assessed by Visual Analogue Scale（VAS）,(0,no pain；10，the worst pain)
Chest pain at rest | Time3: 6 hours after surgery
  Assessed by Visual Analogue Scale（VAS）,(0,no pain；10，the worst pain)
Chest pain at rest | Time4: 24 hours after surgery
  Assessed by Visual Analogue Scale（VAS）,(0,no pain；10，the worst pain)
Chest pain at rest | Time5: 48 hours after surgery
  Assessed by Visual Analogue Scale（VAS）,(0,no pain；10，the worst pain)
Chest pain during deep breath | Time1:0 minute after the first pain score could be obtained from the patient
  Assessed by Visual Analogue Scale（VAS）,(0,no pain；10，the worst pain)
Chest pain during deep breath | Time2: 3 hours after surgery
  Assessed by Visual Analogue Scale（VAS）,(0,no pain；10，the worst pain)
Chest pain during deep breath | Time3: 6 hours after surgery
  Assessed by Visual Analogue Scale（VAS）,(0,no pain；10，the worst pain)
Chest pain during deep breath | Time4: 24 hours after surgery
  Assessed by Visual Analogue Scale（VAS）,(0,no pain；10，the worst pain)
Chest pain during deep breath | Time5: 48 hours after surgery
  Assessed by Visual Analogue Scale（VAS）,(0,no pain；10，the worst pain)
Ear pain at rest | Time1:0 minute after the first pain score could be obtained from the patient
  Assessed by Visual Analogue Scale（VAS）,(0,no pain；10，the worst pain)
Ear pain at rest | Time2: 3 hours after surgery
  Assessed by Visual Analogue Scale（VAS）,(0,no pain；10，the worst pain)
Ear pain at rest | Time3: 6 hours after surgery
  Assessed by Visual Analogue Scale（VAS）,(0,no pain；10，the worst pain)
Ear pain at rest | Time4: 24 hours after surgery
  Assessed by Visual Analogue Scale（VAS）,(0,no pain；10，the worst pain)
Ear pain at rest | Time5: 48 hours after surgery
  Assessed by Visual Analogue Scale（VAS）,(0,no pain；10，the worst pain)
Ear pain during deep breath | Time1:0 minute after the first pain score could be obtained from the patient
  Assessed by Visual Analogue Scale（VAS）,(0,no pain；10，the worst pain)
Ear pain during deep breath | Time2: 3 hours after surgery
  Assessed by Visual Analogue Scale（VAS）,(0,no pain；10，the worst pain)
Ear pain during deep breath | Time3: 6 hours after surgery
  Assessed by Visual Analogue Scale（VAS）,(0,no pain；10，the worst pain)
Ear pain during deep breath | Time4: 24 hours after surgery
  Assessed by Visual Analogue Scale（VAS）,(0,no pain；10，the worst pain)
Ear pain during deep breath | Time5: 48 hours after surgery
  Assessed by Visual Analogue Scale（VAS）,(0,no pain；10，the worst pain)
PCIA consumption | Time1:3 hours after surgery
  Assessed by consumption of patient-controlled intravenous analgesia
PCIA consumption | Time2:6 hours after surgery
  Assessed by consumption of patient-controlled intravenous analgesia
PCIA consumption | Time3:24 hours after surgery
  Assessed by consumption of patient-controlled intravenous analgesia
PCIA consumption | Time4:48 hours after surgery
  Assessed by consumption of patient-controlled intravenous analgesia
Nausea severity | Time1:3 hours after surgery
  Assessed by Verbal Rating Scale（VRS）,(0,no pain；10，the worst pain)
Nausea severity | Time2:6 hours after surgery
  Assessed by Verbal Rating Scale（VRS）,(0,no pain；10，the worst pain)
Nausea severity | Time3:24 hours after surgery
  Assessed by Verbal Rating Scale（VRS）,(0,no pain；10，the worst pain)
Nausea severity | Time4:48 hours after surgery
  Assessed by Verbal Rating Scale（VRS）,(0,no pain；10，the worst pain)
Number of vomiting | Time1:3 hours after surgery
  Assessed by vomiting times after surgery
Number of vomiting | Time2:6 hours after surgery
  Assessed by vomiting times after surgery
Number of vomiting | Time3:24 hours after surgery
  Assessed by vomiting times after surgery
Number of vomiting | Time4:48 hours after surgery
  Assessed by vomiting times after surgery
Intraoperative fentanyl requirement | Time1:0 minute after surgery
  Assessed by total requirement of fentanyl( µg/kg) during the surgery

SECONDARY OUTCOMES:
The first time of urination | Time1:0 minute after the first time of urination
  Assessed by the duration(hour) between end of surgery and the first time of urination
Blood loss during harvesting rib cartilage | Time1:0 minute after all three rib cartilage are harvested
  Assessed by the blood loss(ml)
  ) when surgeons are harvesting rib cartilage for auricular reconstruction
Fentanyl requirement in PACU | Time1:0 minute after departure from the PACU
  Assessed by total additional requirement of fentanyl for keeping VAS scores less than '5'

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Hu, Master, Principal Investigator — Eye and ENT Hospital of Fudan University
Locations (1):
- The Eye,Ear,Nose and throat Hospital ,Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nagata S. A new method of total reconstruction of the auricle for microtia. Plast Reconstr Surg. 1993 Aug;92(2):187-201. doi: 10.1097/00006534-199308000-00001. PMID 8337267
- [Background] Lukosiene L, Rugyte DC, Macas A, Kalibatiene L, Malcius D, Barauskas V. Postoperative pain management in pediatric patients undergoing minimally invasive repair of pectus excavatum: the role of intercostal block. J Pediatr Surg. 2013 Dec;48(12):2425-30. doi: 10.1016/j.jpedsurg.2013.08.016. PMID 24314181
- [Background] Lukosiene L, Macas A, Trepenaitis D, Kalibatiene L, Malcius D, Barauskas V. Single shot intercostal block for pain management in pediatric patients undergoing the Nuss procedure: a double-blind, randomized, controlled study. J Pediatr Surg. 2014 Dec;49(12):1753-7. doi: 10.1016/j.jpedsurg.2014.09.014. Epub 2014 Oct 1. PMID 25487477
- [Background] Willschke H, Marhofer P, Bosenberg A, Johnston S, Wanzel O, Cox SG, Sitzwohl C, Kapral S. Ultrasonography for ilioinguinal/iliohypogastric nerve blocks in children. Br J Anaesth. 2005 Aug;95(2):226-30. doi: 10.1093/bja/aei157. Epub 2005 May 27. PMID 15923270
- [Background] Vemula R, Kutzin M, Greco G, Kutzin T. The use of intercostal nerve blocks for implant-based breast surgery. Plast Reconstr Surg. 2013 Jul;132(1):178e-180e. doi: 10.1097/PRS.0b013e3182911018. No abstract available. PMID 23806943